CLINICAL TRIAL: NCT06172153
Title: Diagnostic Efficacy of Metagenomic Next-generation Sequencing in Patients With Spinal Infections: A Retrospective Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-1095-01
Record Dates: First submitted 2023-12-07; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Spinal Infection; Diagnositic Efficacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sun Yat-sen memorial hospital: Patients who were suspected of Spinal infection.
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No intervention

SUMMARY:
Comparing the diagnostic efficacy between traditional laboratory methods and second-generation high-throughput sequencing in patients suspected of spinal infections.

ELIGIBILITY:
Inclusion Criteria:

"Patients suspected of spinal infections, as per the American Infectious Diseases Society's 2015 criteria for primary vertebral osteomyelitis, were identified based on their clinical symptoms, laboratory tests, and imaging examinations. All cases included in the study underwent laboratory examinations, histopathological examinations, and second-generation high-throughput sequencing (metagenomic sequencing)."

Exclusion Criteria:

"The absence of laboratory examinations, histopathological examinations, and results from second-generation high-throughput sequencing (metagenomic sequencing)."

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: "The patients suspected of spinal infections were admitted to the Orthopedic Department of Sun Yat-sen Memorial Hospital, Sun Yat-sen University."
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
The diagnositic efficacy | 1 year
  Sensitivity, Specificity
The diagnositic efficacy | 1 year
  Positive Predictive Value, Negative Predictive Value

CONTACTS AND LOCATIONS:
Overall Officials: Chunhai Li, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen memorial hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No